CLINICAL TRIAL: NCT00981682
Title: A Phase III Open-Label Extension Study to Investigate the Safety of SER120 Nasal Spray Formulations in Patients With Nocturia Completing Study SPC-SER120-DB1-200901 or Study SPC-SER120-DB2-200902
Brief Title: Long Term Safety Assessment of SER120 in Patients With Nocturia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serenity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPC-SER120-OL1-200903
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2014-01

CONDITIONS: Nocturia
Keywords: decrease in the number of nocturic episodes for patients with nocturia
MeSH Terms: conditions — Nocturia

ARMS (1):
- SER120 (desmopressin) (Experimental)
  Interventions: Drug: SER120

INTERVENTIONS:
Drug: SER120 — once a day treatment of nocturia

SUMMARY:
The hypothesis of this study is that SER120 is safe and well tolerated for use in nocturic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients completed SPC-SER120-DB1-200901 and SPC-SER120-DB2-200902 studies
* Willing to provide consent for the study

Exclusion Criteria:

* Incontinence
* Diabetes Insipidus, Diabetes Mellitus
* CHF
* Renal Insufficiency
* Significant medical history which make participation unacceptable

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stephen M. Auerbach, MD, Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SER120 750 mcg: All participants received up to 750 mcg SER120 once daily
Period: Overall Study
Arm/Group | SER120 750 mcg
Started | 376
Completed | 234
Not Completed | 142
Not completed — Adverse Event | 48
Not completed — Withdrawal by Subject | 52
Not completed — Lost to Follow-up | 14
Not completed — Lack of Efficacy | 13
Not completed — Protocol Violation | 6
Not completed — administrative | 9

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | SER120 750 mcg
Number analyzed (Participants) | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 250
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 376

OUTCOME MEASURES:

1. Primary Outcome: Mean Serum Sodium
Description: Change in mean serum sodium on Day 8, Day 15, Day 22, Week 4, Week 8, Week 12, Week 20, Week 28 and Week 40 compared to Baseline
Time Frame: 40 weeks
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SER120 750 mcg
Number analyzed (Participants) | 376
mmol/L
  Day 8 | -0.0 (2.3)
  Day 15 | -0.4 (2.3)
  Day 22 | -0.4 (2.5)
  Week 4 | -0.3 (2.2)
  Week 12 | -0.5 (2.6)
  Week 20 | -0.4 (2.6)
  Week 28 | -0.8 (2.4)
  Week 40 | -0.6 (2.6)

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | SER120 750 mcg
All-Cause Mortality (participants affected / at risk) | 30/376
Serious Adverse Events (participants affected / at risk) | 30/376
Other Adverse Events (participants affected / at risk) | 305/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 750 mcg (N=376)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Cardiovascular disorders (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
pericarditis (Cardiac disorders) | 1 (1)
sick sinus syndrome (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
overdose (Injury, poisoning and procedural complications) | 1 (1)
post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
alcoholism (Psychiatric disorders) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
gastric banding (Surgical and medical procedures) | 1 (1)
medical device removal (Surgical and medical procedures) | 1 (1)
Uvulopalatopharyngoplasty (Surgical and medical procedures) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SER120 750 mcg (N=376)
Upper respiratory infection (Infections and infestations) | 23 (23)
Nasopharyngitis (Infections and infestations) | 20 (20)
sinusitis (Infections and infestations) | 17 (17)
headache (Nervous system disorders) | 33 (33)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 86 (86)
sneezing (Respiratory, thoracic and mediastinal disorders) | 46 (46)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 43 (43)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (19)
cough (Respiratory, thoracic and mediastinal disorders) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No